CLINICAL TRIAL: NCT04983043
Title: A Multi-center, Randomized, Double-blind, Placebo-parallel Controlled, Standardise-loaded Ⅱ Clinical Trial of Efficacy and Safety of QiShen YiQi Dripping Pills in Chronic Heart Failure
Brief Title: Efficacy and Safety of QiShen YiQi Dripping Pills in Chronic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-QSYQDW-HFrEF-Ⅱ
Record Dates: First submitted 2021-07-08; First posted 2021-07-30 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-03

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): Low dose QiShen YiQi Dripping Pills, 3 bags, take orally after meals, 3 times a day
  Interventions: Drug: Low dose QiShen YiQi Dripping Pills 3 bags
- High dose group (Experimental): High dose QiShen YiQi Dripping Pills, 3 bags, take orally after meals, 3 times a day
  Interventions: Drug: High dose QiShen YiQi Dripping Pills 3 bags
- Placebo group (Placebo Comparator): QiShen YiQi Dripping Pills placebo, 3 bags, take orally after meals, 3 times a day
  Interventions: Drug: QiShen YiQi Dripping Pills placebo 3 bags

INTERVENTIONS:
Drug: Low dose QiShen YiQi Dripping Pills 3 bags — Low dose QiShen YiQi Dripping Pills contain QiShen YiQi Dripping Pills 2 bags(0.52g dripping pills per bag) and QiShen YiQi Dripping Pills placebo 1 bag(0.52g dripping pills placebo per bag),take orally after meals, 3 times a day for 12weeks
  Other Names: Low dose group
  Arms: Low dose group
Drug: High dose QiShen YiQi Dripping Pills 3 bags — High dose QiShen YiQi Dripping Pills contain QiShen YiQi Dripping Pills 3 bags(0.52g dripping pills per bag),take orally after meals, 3 times a day for 12weeks
  Other Names: High dose group
  Arms: High dose group
Drug: QiShen YiQi Dripping Pills placebo 3 bags — QiShen YiQi Dripping Pills placebo contain QiShen YiQi Dripping Pills placebo 3 bags(0.52g dripping pills placebo per bag),take orally after meals, 3 times a day for 12weeks
  Other Names: Placebo group
  Arms: Placebo group

SUMMARY:
This study will evaluate the efficacy and safety and the best effective dose of QiShen YiQi Dripping Pills in the treatment of chronic heart failure with decreased ejection fraction of CHD (Qi deficiency and blood stasis syndrome).

DETAILED DESCRIPTION:
QiShen YiQi Dripping Pills are oral, compound traditional chinese medicine prepatations. This study will evaluate the efficacy and safety and the best effective dose of QiShen YiQi Dripping Pills in the treatment of chronic heart failure with decreased ejection fraction of CHD (Qi deficiency and blood stasis syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Conformed to the diagnostic criteria of CHD and chronic heart failure
* Conformed to the TCM syndrome differentiation standard of chronic heart failure syndrome of Qi deficiency and blood stasis
* Male or female subjects aged ≥ 40 years and ≤80 years
* LVEF<45%(modified Simpson method)
* NYHAⅡ-Ⅲ
* Received standardized drug therapy for chronic heart failure at least 2 weeks before randomization, and did not receive intravenous therapy (vasoactive drugs, diuretics) within 2 weeks without adjustment of dose
* Ability to understand the requirements of the study and willingness to provide written informed consent
* Have no pregnancy program and take effective contraceptive measures voluntarily
* Abide by the experimental protocol and cooperate with the data collection according to the researcher's judgment

Exclusion Criteria:

* Patients with heart failure caused by other heart diseases,such as cor pulmonale, congenital heart disease, primary pulmonary hypertension, secondary severe pulmonary hypertension, severe stenosis or insufficiency of heart valves, cardiomyopathy (including hypertrophic cardiomyopathy, restrictive cardiomyopathy, dilated cardiomyopathy, alcoholic cardiomyopathy), moderate massive pericardial effusion, constrictive pericarditis, infective endocarditis
* Heart failure caused by systemic diseases or other systemic diseases, such as rheumatic immune and secretory diseases;heart failure caused by kidney disease, lung disease, liver disease and serious infection;heart failure caused by chemical or toxicological causes
* Patients who had acute myocardial infarction, underwent coronary revascularization or left ventricular remodeling, underwent cardiac resynchronization with pacemaker implantation, underwent cardiothoracic surgery within 3 months prior to receiving the experimental drug, patients with other acute coronary syndrome, pulmonary embolism or acute cerebrovascular disease
* Severe arrhythmias such as ventricular tachycardia, second degree Ⅱ type or above sinus atrial or atrioventricular block without pacemaker treatment, average QTc > 500ms, heart rate < 50 beats/min, etc
* Complicated with other serious diseases, such as pheochromocytoma, hematologic diseases, organ transplantation patients, and any history of malignant tumor
* The presence of uncontrolled hypertension, systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg
* Hypotension with a systolic blood pressure <80mmHg and/or a diastolic blood pressure <50mmHg
* Patients with hepatic and/or renal dysfunction (ALT≥ 2 times the upper limit of normal, and/or estimated glomerular filtration rate (EGFR) <30 mL /min/1.73m2
* HbA1c ≥9.0%, or fasting blood glucose ≥13.9mmol/L
* Moderate and severe anemia (Hb < 90g/L)
* Serum potassium ≥5.5mmol/L
* Patients requiring anticoagulants who did not achieve dose stabilization for 1 month or INR > 3.0
* In patients who need to take antiplatelet drugs, the dose was stable for less than 1 month, and the platelet value was lower than the lower limit of normal value
* Allergic to the test drug or its related taste or ingredients
* People with complicated mental illness, poor condition control and drug addiction
* Unable to complete 6MWT
* Pregnant or lactating women
* Participation in other studies and use of investigational drugs from other studies within 3 months prior to screening
* The investigator deems that the patient is not suitable to participate in the study, including the investigator's judgment that the patient is unable to complete the study or comply with the requirements of the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
6-Minutes-Walking-Test (6MWT) in week 12 | Baseline to weeks 12
  Change from baseline to weeks 12 in exercise capacity as measured by the 6-Minutes-Walking-Test (6MWT) distance.

SECONDARY OUTCOMES:
6-Minutes-Walking-Test (6MWT) in weeks 4 and 8 | Baseline to weeks 4 and 8
  Change from baseline to weeks 4 and 8 in exercise capacity as measured by the 6-Minutes-Walking-Test (6MWT) distance.
NYHA classification | Baseline to weeks 4,8 and 12
  Percentage of subjects whose NYHA classification improved/worsened/remained unchanged from baseline to weeks 4,8 and 12.
Traditional Chinese Medicine Syndrome Score | Baseline to weeks 4,8 and 12
  Change from baseline to weeks 4,8 and 12 in Traditional Chinese Medicine Syndrome Score. There were 3 clinical primary symptoms, 4 clinical secondary symptoms, tongue picture and pulse condition evaluated as TCM symptoms, which was defined as TCM syndrome score. The standard of TCM primary symptoms scored as without 0, light 2, medium 4, heavy 6 points. The standard of TCM secondary symptoms scored as without 0, with 1 points. Tongue picture and pulse condition did not count.
Dyspnea, weakness, edema | Baseline to weeks 4,8 and 12
  Symptom disappearance rate(dyspnea, weakness, edema) from baseline to weeks 4,8 and 12.
Echocardiogram results | Baseline to weeks 4,8 and 12
  1. Change from baseline to weeks 4,8 and 12 in left ventricular end diastolic diameter(LVEDD) measured by echocardiography;
  2. Change from baseline to weeks 4,8 and 12 in left ventricular end diastolic volume(LVEDV) measured by echocardiography;
  3. Change from baseline to weeks 4,8 and 12 in left ventricular end systolic volume(LVESV) measured by echocardiography;
  4. Change from baseline to weeks 4,8 and 12 in left ventricular ejection fraction(LVEF) measured by echocardiography;
  5. Change from baseline to weeks 4,8 and 12 in stroke volume(SV) measured by echocardiography;
  6. Change from baseline to weeks 4,8 and 12 in cardiac output(CO) measured by echocardiography.
NT-proBNP | Baseline to weeks 4,8 and 12
  Change from baseline to weeks 4,8 and 12 in NT-proBNP.
Minnesota Living With Heart Failure Questionnaire(MLHFQ) | Baseline to weeks 4,8 and 12
  Change from baseline to weeks 4,8 and 12 in Minnesota Living With Heart Failure Questionnaire(MLHFQ). The MLHFQ is a self-administered questionnaire for patients with HF, comprising 21 items representing different degrees of impact of HF on health-related quality of life. Every item in this questionnaire scores from 0 (none) to 5 (very much) and the total items score from 0 (none) to 105 (very much).
Cardiovascular adverse events | Week 12
  To determine whether the incidence of cardiovascular adverse events during the study period was superior to placebo.

OTHER OUTCOMES:
Saturation of Peripheral Oxygen | Week 12
  To determine whether the saturation of peripheral oxygen is improved from baseline to week 12 after treatment.
Grasp strength body mass index test | Week 12
  To determine whether the grasp strength body mass index is improved from baseline to week 12 after treatment.

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Hefei First People's Hospital, Hefei, Anhui
  - The First Hospital of ANHUI University of Science & Technology, Huainan, Anhui
  - Suzhou Municipal Hospital, Suzhou, Anhui
  - Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - Dongguan TCM Hospital, Dongguan, Guangdong
  - Nanfang Hospital，Southern Medical University, Guangzhou, Guangdong
  - The Affiliated TCM Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Zhong Shan Hospital of Chinese Medicine, Zhongshan, Guangdong
  - Ruikang Hospital Affiliated to Guangxi University of Traditional Chinese Medicine, Nanning, Guangxi
  - The First Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Luoyang Third People's Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Pepole's Hospital of Xinzheng, Zhengzhou, Henan
  - Hunan University of Chinese Medicine, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Nanjing Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - The Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Xi'an Daxing Hospital, Xi'an, Shaanxi
  - The Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - The Second Affiliated Hospital of Tianjin University of traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Hospital of Traditional Chinese Medicine of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang

REFERENCES:
- [Derived] He X, Jiang Y, Li S, Liu D, Li Z, Han X, Zhang X, Dong X, Liu H, Huang J, Wang X, Long W, Ni S, Yang Z, Ye T. Efficacy and Safety of QiShen YiQi Dripping Pills in the Treatment of Coronary Heart Disease Complicating Chronic Heart Failure (Syndrome of Qi Deficiency with Blood Stasis): Study Protocol for a Randomized, Placebo-Controlled, Double-Blind and Multi-Centre Phase II Clinical Trial. Int J Gen Med. 2023 Dec 28;16:6177-6188. doi: 10.2147/IJGM.S436999. eCollection 2023. PMID 38169574